CLINICAL TRIAL: NCT06860295
Title: The Architectural Immunoregulation in Atherosclerotic Disease: A Single-Cell RNA Sequencing and Spatial Biology Approach
Brief Title: "Immunoregulation in Atherosclerosis: A Single-Cell RNA Sequencing Study"
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Principal Investigator, Carlos Vicente Serrano Junior, Principal Investigator, Hospital Israelita Albert Einstein
Other Study IDs: AteroImunoHIAE
Record Dates: First submitted 2025-02-24; First posted 2025-03-06 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Atherosclerosis of Coronary Artery
Keywords: Atherosclerosis; Single Cell RNA-sequencing; Immunology
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Tissue Dissociation
  The tissue from the plates will be enzymatically dissociated into single-cell suspensions using a combination of collagenase, DNase I, and dispase.
  Cells will be filtered through a 70 µm filter to remove debris and aggregates. Viability Check and Enrichment
  Cell viability will be assessed using Trypan blue exclusion. Dead cells and debris will be removed using a magnetic kit for dead cell removal, if necessary.
  scRNAseq Workflow Library Preparation
  Single-cell capture and library preparation will be performed using a droplet-based microfluidic system (e.g., 10x Genomics Chromium).
  Approximately 5,000-10,000 cells per sample will be targeted for analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Coronary Plaques from Explanted Heart: The selected arteries will be dissected and microscopically evaluated, and the samples will be fixed in formalin, embedded in paraffin, and stained for histological analysis. The tissue will be enzymatically dissociated to obtain individual cells, which will then be filtered and assessed for cell viability. The cells will undergo single-cell RNA sequencing (scRNAseq) with the aim of analyzing around 5,000-10,000 cells per sample. The sample size will be 20-30 plaques, with the goal of capturing the main cellular populations and performing a robust analysis.
  Interventions: Diagnostic Test: Single Cell RNA Sequencing

INTERVENTIONS:
Diagnostic Test: Single Cell RNA Sequencing — Reprocessing
  Data normalization, dimensionality reduction, and clustering will be performed using the Seurat package (based on R).
  Cell types will be identified based on canonical marker gene expression. Cell Subpopulation Identification
  Clusters will be annotated based on signatures of known cell types (e.g., endothelial cells, smooth muscle cells, macrophages, etc.).
  Differential gene expression analysis will be conducted to identify disease-associated genes.
  Pathway and Function Enrichment
  Gene Set Enrichment Analysis (GSEA) and pathway analyses (e.g., KEGG, Reactome) will be carried out to investigate the biological processes and pathways driving atherosclerosis.
  Quality Control
  Sequencing reads will be assessed for quality using FASTQC, and low-quality reads will be filtered out.
  The Cell Ranger software (10x Genomics) will be used to align reads to the human genome and quantify gene expression at the single-cell level.

SUMMARY:
Atherosclerosis is the leading cause of acute cardiovascular events, such as myocardial infarction and stroke, and is a significant risk factor for cardiovascular mortality. The detailed understanding of the immune mechanisms and cellular transformations involved in the pathogenesis of atherosclerosis is still limited, and the use of single-cell RNA sequencing (scRNAseq) has revealed new cellular functions and subpopulations associated with disease progression. This study aims to identify cellular subpopulations, molecular pathways, and changes in gene expression related to the development of atherosclerosis in human coronary arteries. Using scRNAseq, the study seeks to characterize the transcriptomic landscape of cells present in atherosclerotic plaques and identify molecular signatures that reveal individual predispositions to specific phenotypes, such as disease susceptibility and response to therapies. The research will be conducted at the Albert Einstein Israeli Hospital in São Paulo and will involve samples from coronary arteries and atherosclerotic plaques of the explanted hearts of patients who have undergone heart transplants as well as from discarded material of coronary artery bypass graft surgery (CABG). With an estimated sample size of 20-30 plaques, the data obtained will allow for a detailed analysis of the molecular mechanisms involved in atherosclerosis, contributing to the development of specific therapeutic targets.

DETAILED DESCRIPTION:
This is a prospective observational study that will be conducted with samples of coronary arteries and atherosclerotic plaques from the explanted hearts of patients with ischemic cardiomyopathy who have undergone heart transplants as well as from discarded material of coronary artery bypass graft surgery . The atherosclerotic plaque samples will be retrieved from the coronary arteries during the transplant surgery or the CABG procedure and transported to the laboratory within 2 hours. The selected arteries will be dissected and microscopically evaluated, and the samples will be fixed in formalin, embedded in paraffin, and stained for histological analysis. The tissue will be enzymatically dissociated to obtain individual cells, which will then be filtered and assessed for cell viability. The cells will undergo single-cell RNA sequencing (scRNAseq) with the aim of analyzing around 5,000-10,000 cells per sample. The sample size will be 20-30 plaques, with the goal of capturing the main cellular populations and performing a robust analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with ischemic cardiomyopathy due to advanced atherosclerosis, undergoing heart transplantation;
* Patients with coronary artery disease submitted to coronary artery bypass graft surgery (CABG)."
* Aged between 40 and 75 years;
* Signed informed consent form.

Exclusion Criteria:

* Patients with systemic inflammatory or autoimmune diseases;
* History of cancer within the last 5 years or active malignancy;
* Recent use (within the last 6 months) of immunosuppressive therapy.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with ischemic cardiomyopathy due to advanced atherosclerosis, undergoing heart transplantation.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-06-25 (Estimated); Primary Completion 2026-10-25 (Estimated); Study Completion 2027-04-25 (Estimated)

PRIMARY OUTCOMES:
Concentration of Specific Cells Clusters And Macrophage / Linfocite Subpopulations : Create a high-resolution single-cell atlas of atherosclerotic plaques. | Through study completion, an average of 1 year and a half.
  Determine the concentration of cellular clusters with specific inflammatory subpopulations determination to Create a high-resolution single-cell atlas of atherosclerotic plaques, revealing cell-specific transcriptional changes associated with the disease. The findings could identify new therapeutic targets for intervention in atherosclerosis and enhance the understanding of its molecular pathogenesis.

SECONDARY OUTCOMES:
Concentration of interleukins and cellular subtypes by citometer flow to Identification of molecular signatures in atherosclerosis | Through study completion, an average of 1 year and a half .
  The secondary objective is to identify molecular signatures that reveal individual predispositions to specific phenotypes, such as susceptibility to atherosclerosis, response to therapies, and other health characteristics, establishing the foundation for precision medicine and population health studies in Brazil by determining specific concentrations of pro and anti-inflammatory molecules and cell types.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The scRNA-seq data and R scripts used in the analysis of this study will be available from the corresponding author upon request.
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Background] Zhang H, Viveiros A, Nikhanj A, Nguyen Q, Wang K, Wang W, Freed DH, Mullen JC, MacArthur R, Kim DH, Tymchak W, Sergi CM, Kassiri Z, Wang S, Oudit GY. The Human Explanted Heart Program: A translational bridge for cardiovascular medicine. Biochim Biophys Acta Mol Basis Dis. 2021 Jan 1;1867(1):165995. doi: 10.1016/j.bbadis.2020.165995. Epub 2020 Oct 22. PMID 33141063
- [Background] Rajab TK, Singh SK. Donation After Cardiac Death Heart Transplantation in America Is Clinically Necessary and Ethically Justified. Circ Heart Fail. 2018 Mar;11(3):e004884. doi: 10.1161/CIRCHEARTFAILURE.118.004884. No abstract available. PMID 29664408
- [Background] Price AL, Patterson N, Yu F, Cox DR, Waliszewska A, McDonald GJ, Tandon A, Schirmer C, Neubauer J, Bedoya G, Duque C, Villegas A, Bortolini MC, Salzano FM, Gallo C, Mazzotti G, Tello-Ruiz M, Riba L, Aguilar-Salinas CA, Canizales-Quinteros S, Menjivar M, Klitz W, Henderson B, Haiman CA, Winkler C, Tusie-Luna T, Ruiz-Linares A, Reich D. A genomewide admixture map for Latino populations. Am J Hum Genet. 2007 Jun;80(6):1024-36. doi: 10.1086/518313. Epub 2007 Apr 13. PMID 17503322
- [Background] Gouveia MH, Bentley AR, Leal TP, Tarazona-Santos E, Bustamante CD, Adeyemo AA, Rotimi CN, Shriner D. Unappreciated subcontinental admixture in Europeans and European Americans and implications for genetic epidemiology studies. Nat Commun. 2023 Nov 7;14(1):6802. doi: 10.1038/s41467-023-42491-0. PMID 37935687
- [Background] Hu Z, Liu W, Hua X, Chen X, Chang Y, Hu Y, Xu Z, Song J. Single-Cell Transcriptomic Atlas of Different Human Cardiac Arteries Identifies Cell Types Associated With Vascular Physiology. Arterioscler Thromb Vasc Biol. 2021 Apr;41(4):1408-1427. doi: 10.1161/ATVBAHA.120.315373. Epub 2021 Feb 25. PMID 33626908
- [Background] Soehnlein O, Libby P. Targeting inflammation in atherosclerosis - from experimental insights to the clinic. Nat Rev Drug Discov. 2021 Aug;20(8):589-610. doi: 10.1038/s41573-021-00198-1. Epub 2021 May 11. PMID 33976384
- [Background] Fernandez DM, Rahman AH, Fernandez NF, Chudnovskiy A, Amir ED, Amadori L, Khan NS, Wong CK, Shamailova R, Hill CA, Wang Z, Remark R, Li JR, Pina C, Faries C, Awad AJ, Moss N, Bjorkegren JLM, Kim-Schulze S, Gnjatic S, Ma'ayan A, Mocco J, Faries P, Merad M, Giannarelli C. Single-cell immune landscape of human atherosclerotic plaques. Nat Med. 2019 Oct;25(10):1576-1588. doi: 10.1038/s41591-019-0590-4. Epub 2019 Oct 7. PMID 31591603
- [Background] Wirka RC, Wagh D, Paik DT, Pjanic M, Nguyen T, Miller CL, Kundu R, Nagao M, Coller J, Koyano TK, Fong R, Woo YJ, Liu B, Montgomery SB, Wu JC, Zhu K, Chang R, Alamprese M, Tallquist MD, Kim JB, Quertermous T. Atheroprotective roles of smooth muscle cell phenotypic modulation and the TCF21 disease gene as revealed by single-cell analysis. Nat Med. 2019 Aug;25(8):1280-1289. doi: 10.1038/s41591-019-0512-5. Epub 2019 Jul 29. PMID 31359001
- [Background] Kim K, Park SE, Park JS, Choi JH. Characteristics of plaque lipid-associated macrophages and their possible roles in the pathogenesis of atherosclerosis. Curr Opin Lipidol. 2022 Oct 1;33(5):283-288. doi: 10.1097/MOL.0000000000000842. Epub 2022 Aug 3. PMID 35942822
- [Background] Chattopadhyay A, Guan P, Majumder S, Kaw K, Zhou Z, Zhang C, Prakash SK, Kaw A, Buja LM, Kwartler CS, Milewicz DM. Preventing Cholesterol-Induced Perk (Protein Kinase RNA-Like Endoplasmic Reticulum Kinase) Signaling in Smooth Muscle Cells Blocks Atherosclerotic Plaque Formation. Arterioscler Thromb Vasc Biol. 2022 Aug;42(8):1005-1022. doi: 10.1161/ATVBAHA.121.317451. Epub 2022 Jun 16. PMID 35708026
- [Background] Su C, Lu Y, Wang Z, Guo J, Hou Y, Wang X, Qin Z, Gao J, Sun Z, Dai Y, Liu Y, Liu G, Xian X, Cui X, Zhang J, Tang J. Atherosclerosis: The Involvement of Immunity, Cytokines and Cells in Pathogenesis, and Potential Novel Therapeutics. Aging Dis. 2023 Aug 1;14(4):1214-1242. doi: 10.14336/AD.2022.1208. PMID 37163428
- [Background] Serrano CV Jr, Yoshida VM, Venturinelli ML, D'Amico E, Monteiro HP, Ramires JA, da Luz PL. Effect of simvastatin on monocyte adhesion molecule expression in patients with hypercholesterolemia. Atherosclerosis. 2001 Aug;157(2):505-12. doi: 10.1016/s0021-9150(00)00757-7. PMID 11472753
- [Background] Li Q, Wang M, Zhang S, Jin M, Chen R, Luo Y, Sun X. Single-cell RNA sequencing in atherosclerosis: Mechanism and precision medicine. Front Pharmacol. 2022 Oct 4;13:977490. doi: 10.3389/fphar.2022.977490. eCollection 2022. PMID 36267275
- [Background] Serrano CV Jr, de Mattos FR, Pitta FG, Nomura CH, de Lemos J, Ramires JAF, Kalil-Filho R. Association between Neutrophil-Lymphocyte and Platelet-Lymphocyte Ratios and Coronary Artery Calcification Score among Asymptomatic Patients: Data from a Cross-Sectional Study. Mediators Inflamm. 2019 Mar 26;2019:6513847. doi: 10.1155/2019/6513847. eCollection 2019. PMID 31049026
- [Background] Makover ME, Shapiro MD, Toth PP. There is urgent need to treat atherosclerotic cardiovascular disease risk earlier, more intensively, and with greater precision: A review of current practice and recommendations for improved effectiveness. Am J Prev Cardiol. 2022 Aug 6;12:100371. doi: 10.1016/j.ajpc.2022.100371. eCollection 2022 Dec. PMID 36124049